CLINICAL TRIAL: NCT00829036
Title: Wayfinding Information Access System for People With Vision Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: C6690-R
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-02

CONDITIONS: Blindness
Keywords: Rehabilitation; Sensory Aid
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Wayfinding Prototype (Experimental): A Wayfinding Prototype is evaluated in terms of the time it takes subjects to use this device to walk to specific indoor locations versus baseline walking time.
  Interventions: Device: Wayfinding Prototype

INTERVENTIONS:
Device: Wayfinding Prototype — A Wayfinding Prototype is used by subjects to determine any advantages over current standard of rehabilitation.

SUMMARY:
The purpose of the project is to find out what kinds of information are most useful to visually impaired people when they are moving around indoors and what kinds of controls will make it easy for visually impaired people to control a device to help orient them to an unfamiliar indoor space.

DETAILED DESCRIPTION:
The greatest mobility problems for people with severe visual impairment are caused by gaps in available information about the environment -- environmental cues needed for orienting to salient landmarks in the surrounding environment and for wayfinding. Such informational cues are of great import because persons with severe visual impairment can become hopelessly lost if they cannot keep track of where they are at any given moment as they move along.

A newly developed long-range Radio Frequency Identification (RFID) tag reader might completely solve this problem. Previously, passive (i.e., not battery powered) RFID tags could only be read from a distance of 16 inches or less. This new tag reader can read multiple tags up to 18 feet away, and indicate the direction and range of each tag. At a cost of under 10 each, 250 RFID tags would have to be placed around an environment to equal the cost of 1 Braille sign ($25), yet the value-added in terms of available information at a distance is incredible: every object (landmark, door, water fountain, exit sign, chair, table, etc.) within a range of 18 feet would be able to "announce" its presence.

Visible signage equivalency could be achieved overnight. Further, Interface, Inc., a commercial floor manufacturer is now adhering RFID tags to the protected underside their 50X50 cm floor tiles. Using such flooring and the new long-range readers, a very elegant and affordable indoor GPS-like guidance system can be realized through triangulation of these RFID floor tiles. In the long run, as this RFID flooring infrastructure fills in, the most ideal solution could result, as it would enable the development of easily-managed building databases containing everything users would need to know to orient to new buildings and find their way around with ease. Users would never be lost, as they would always know their current location and heading. In addition, such a building database would be much easier to maintain, as opposed to updating individual RFID tags, when building tenants move or renovations take place. Interface is very interested in supporting our research, and is donating 2500 square feet of their RFID flooring to the VA for this purpose.

The Research Questions to be answered by the herein proposed research are:

1. How should environmental information be organized and parsed according to actual needs so that persons can be provided with needed information without inundating them with useless and/or distracting information in the process?
2. How should a user interface be structured to offer needed information in an easily controlled and useable fashion?

To address these Questions, the following Research Objectives have been established:

1. Determine what kinds of information are needed according to (a) a characterization of individual needs, O&M abilities, and degree of useful residual vision;
2. Develop a structured database of information parsed and organized according to information associated with specific participant characterization clusters as associated with individual needs, residual vision, etc.;
3. Develop an optimal user interface for the control and delivery of needed information adaptable to the individual needs of the participants;
4. Develop an RFID reader antenna that can triangulate RFID tags in flooring to determine the user's current location and heading, as well as identify the information and location of other tags of interest on objects in the surround; and
5. Construct and Evaluate a Wayfinding Prototype as specified by the results of the above objectives.

ELIGIBILITY:
Inclusion Criteria:

* Must be blind with no better vision than light perception and must be able to do 3 hours of walking (with many breaks)

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Ross, MSEE Med, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Prototype vs. Baseline: Prototype:
  Subjects are trained for 20 minutes in the use of the prototype (1) in open spaces and (2) in hallways. They are taught how to select a destination, and obtain turn-by-turn navigation directions to walk to the selected destination. Subjects are then asked to walk to 12 different unknown locations, one location in each of 12 timed trials. Half of these locations are in open spaces and half in hallways. Walking time is the performance measure.
  Baseline:
  An Orientation and Mobility (O&M) specialist first teaches the subject how to find (walk to) each of the same 12 locations, though in a different order. Again, 6 of these are in open spaces and 6 in hallways. Then, over 12 trials, subjects are asked to independently walk to each of the specified locations, one location per trial. Again, walking time is the performance measure.
Period: Overall Study
Arm/Group | Prototype vs. Baseline
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Using Repeated Measures ANOVA for the 24 participants, and assuming a minimum correlation between repeated measures of .7, our analyses will be sensitive to a between factor effect size of f=.33, with power set to .80 and alpha level set to .05. This should be sufficient to reveal significant differences between baseline and device use.
Groups:
- Baseline Wayfinding Performance: An Orientation and Mobility specialist teaches subjects (1) how to find each of 4 specific locations in an open space from a random starting location, and (2) how to navigate hallways from a known starting location to find each of 8 specific locations in the hallways of the Atlanta VA Medical Center. Subjects are then (1) brought to a random start point in the open space and asked to walk to the same 4 specific locations they were taught to find and (2) brought to a known starting point in the hallways of the VA Medical Center and asked to walk to the same 8 specific locations they were taught to find.
Arm/Group | Baseline Wayfinding Performance
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 14
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent (Prototype / Baseline) Time
Description: The outcome measure for each subject is the mean of the (Prototype Time / Baseline Time) across 12 trials. The outcome measure for the experiment is the mean of 24 individual subject mean scores. This mean outcome measure is expressed as a percentage of the mean Baseline Time, where improved performance is represented by a percentage that is less than 100 percent of the Baseline Time. The lower the percentage, the better the performance improvement.
Time Frame: 2 hours
Population: Power Analysis: Using Repeated Measures ANOVA for the 24 participants assuming a minimum correlation between repeated measures of .7, we chose our analyses will be sensitive to a medium between factor effect size of f=.33 with power set to .80 and alpha level set to .05.
Measure: Mean (Standard Deviation); unit: Percentage of Baseline Performance Time
Arm/Group | Prototype vs. Baseline
Number analyzed (Participants) | 24
Percentage of Baseline Performance Time | 78.7 (68.6)

ADVERSE EVENTS:
Time Frame: 4 months
Groups:
- Wayfinding: Prototype vs. Baseline: Prototype:
  Subjects are trained to use the prototype to walk to selected destinations (1) in open spaces and (2) through hallways. Then, over 12 trials, subjects are asked to use the prototype to walk to a different unknown location in each trial. Half the locations are in open spaces and half in hallways. Performance time is measured.
  Baseline:
  An Orientation and Mobility (O&M) specialist first teaches the subjects how to find (walk to) 12 specific locations, 6 in open spaces and 6 in hallways. Then, over 12 trials, subjects are asked to independently walk to each of the specified locations. Performance time is measured.
Arm/Group | Wayfinding: Prototype vs. Baseline
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No